CLINICAL TRIAL: NCT01644799
Title: A Phase I Trial of Lenalidomide and Idelalisib in Recurrent Follicular Lymphoma
Brief Title: Lenalidomide and Idelalisib in Treating Patients With Recurrent Follicular Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Gilead Sciences (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A051202; CDR0000736814 (Registry Identifier: PDQ (Physician Data Query)); NCI-2012-01988 (Registry Identifier: CTRP (Clinical Trials Reporting System)); U10CA031946 (NIH)
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Recurrent Follicular Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — idelalisib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lenalidomide and idelalisib (Experimental): Lenalidomide:
  Lenalidomide will be administered orally on days 1-21 followed by 7 days of rest, every 28 days. A treatment cycle will be considered 28 days in length. In the absence of intolerable toxicity or disease progression, lenalidomide will be given for a total of 12 cycles.
  Idelalisib:
  Dosing is fixed in all cohorts receiving idelalisib at 150 mg orally (twice daily) for 12 cycles, with the exception of dose modifications for toxicity.
  Interventions: Drug: idelalisib; Drug: lenalidomide

INTERVENTIONS:
Drug: idelalisib — oral
Drug: lenalidomide — oral

SUMMARY:
Biologic therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Idelalisib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. This phase I trial studies the side effects and the best dose of lenalidomide when giving together with idelalisib in treating patients with recurrent follicular lymphoma.

DETAILED DESCRIPTION:
OUTLINE:

This is a multicenter, dose-escalation study of lenalidomide.

Patients receive lenalidomide orally (PO) on days 1-21 and idelalisib twice daily (BID) on days 1-28. Treatment with lenalidomide and idelalisib repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. The primary and secondary objectives of the study include the following:

Primary Objective:

* To determine the maximum-tolerated dose (MTD) of lenalidomide when combined with idelalisib in patients with recurrent follicular non-Hodgkin lymphoma (NHL).

Secondary Objectives:

* To determine the toxicity profile of lenalidomide and idelalisib therapy in patients with recurrent follicular NHL
* To estimate the efficacy (overall response rate [ORR], complete response rate [CRR], and progression-free survival [PFS]) of lenalidomide and idelalisib in patients with recurrent follicular NHL in a preliminary fashion (using a small extension cohort)
* To assess whether the therapeutic effects of the lenalidomide and idelalisib combination are sufficiently promising to warrant evaluation in a subsequent (phase II/III) randomized trial

After completion of study treatment, patients are followed at 2, 4, 6, 9, 12, 15, 18, and 24 months and then annually. Patients are followed once every year for a maximum of 10 years from study entry.

ELIGIBILITY:
* Documentation of Disease

  * Previously treated, histologically confirmed follicle center cell lymphoma, World Health Organization (WHO) classification grade 1, 2, or 3a (> 15 centroblasts per high-power field with centrocytes present)
  * Bone marrow biopsies as the sole means of diagnosis are not acceptable; fine-needle aspirates are not acceptable for diagnosis
  * Confirmed Cluster of Differentiation 20 (CD20) antigen expression by flow cytometry or immunohistochemistry
* Measurable disease must be > 1 cm
* Prior treatment

  * Patient must have had prior treatment with rituximab either alone or in combination with chemotherapy.
  * Last prior treatment regimen need not include rituximab.
  * Patient must have a time to progression of ≥ 6 months from last rituximab dose of last rituximab containing regimen.
  * No corticosteroids within two weeks prior to study, except for maintenance therapy for a non-malignant disease; maintenance therapy dose may not exceed 20 mg/day prednisone or equivalent
* Patients must be 18 years of age or older.
* Human immunodeficiency virus (HIV) Infection

  * Patients with HIV infection are eligible, provided they meet the following:
  * CD4+ cell count > 350/mm^3
  * Treatment sensitive HIV and, if on anti-HIV therapy, HIV viral load < 50 copies/mm^3
  * No history of Acquired Immunodeficiency Syndrome (AIDS)-defining conditions or other HIV related illness
  * No concurrent zidovudine or stavudine because of overlapping toxicities with protocol therapy
* Patients must not have known central nervous system (CNS) involvement
* Patients must not have known positivity for hepatitis B, as evidenced by + HBsAG or anti-HBc and must not have known history of hepatitis C
* Patients must not have any currently active secondary malignancy except non-melanoma skin cancer. Patients are not considered to have a "currently active" secondary malignancy if they have completed anticancer therapy and are deemed to have < 30% risk of relapse by their physician.
* Patients must not have had deep vein thrombosis or pulmonary embolism within the past 3 months.
* Patients must not have had radioimmunotherapy within 12 months of study entry.
* Patients must not have other concurrent investigational or commercial agents or therapies for lymphoma.
* Patients must not have current dialysis treatment.
* Patients must be non-pregnant and non-nursing.

  * Females of Child Bearing Potential (FCBP) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal for at least 24 consecutive months (eg, has had menses at any time preceding 24 consecutive months)
  * FCBP must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days prior to registration
  * FCBP must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control

    * One highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide
    * FCBP must also agree to ongoing pregnancy testing
  * Men must agree to use a latex condom during sexual contact with a female of childbearing potential, even if they have had a successful vasectomy
* CYP3A4 Strong Inducers and Inhibitors

  * Patients must not be on strong CYP3A4 inhibitors and/or inducers.
  * Strong inhibitors are prohibited: indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketoconazole, nefazodone
  * Strong inducers are prohibited: carbamazepine, phenobarbital, phenytoin, pioglitazone, rifabutin, rifampin, St. John's Wort, troglitazone
* Required Initial Laboratory Values

  * Absolute neutrophil count (ANC) ≥ 1,000 mm³
  * Total Bilirubin ≤ 2 times upper limit of normal (ULN) (unless due to Gilbert disease or lymphoma)
  * Creatinine ≤ 1.5 times ULN (unless due to lymphoma) OR creatinine clearance (CrCl) ≤ 60 mL/minute
  * Platelet count ≥ 75,000 mm³
  * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
MTD based on the incidence of dose-limiting toxicity (DLT) assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 13 months

SECONDARY OUTCOMES:
Toxicity profile assessed by NCI CTCAE version 4.0 | Up to 10 years
OR rate assessed up to 10 years | Up to 10 years
CR rate assessed up to 10 years | Up to 10 years
PFS assessed up to 10 years | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: John P. Leonard, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (6):
- United States (6):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Weill Medical College of Cornell University, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio

REFERENCES:
- [Derived] Smith SM, Pitcher BN, Jung SH, Bartlett NL, Wagner-Johnston N, Park SI, Richards KL, Cashen AF, Jaslowski A, Smith SE, Cheson BD, Hsi E, Leonard JP. Safety and tolerability of idelalisib, lenalidomide, and rituximab in relapsed and refractory lymphoma: the Alliance for Clinical Trials in Oncology A051201 and A051202 phase 1 trials. Lancet Haematol. 2017 Apr;4(4):e176-e182. doi: 10.1016/S2352-3026(17)30028-5. Epub 2017 Mar 15. PMID 28314699